CLINICAL TRIAL: NCT06406920
Title: Intravascular Clotting Detected in Point-of-care Ultrasound as a Marker of the Timing and Severity of Cardiac Arrest and an Indicator of Futile Resuscitation
Brief Title: Intravascular Clotting (POCUS) - Marker of the Timing and Severity of Cardiac Arrest; Indicator of Futile Resuscitation
Status: Recruiting | Type: Observational
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Other Study IDs: 71-01423/K01/61/643/282/2024
Record Dates: First submitted 2024-03-24; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Cardiac Arrest
Keywords: cardiopulmonary resuscitation CPR; point-of-care ultrasound POCUS; intravascular clotting
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The scientific goals of the project:

1. ultrasound assessment of the incidence of clotting in deep veins in patients after cardiac arrest during resuscitation and after the declaration of death; comparison to the incidence of clotting in the heart cavities
2. comparison of resuscitation results in patients with and without clotting detected in deep veins during resuscitation
3. determining the time from cardiac arrest to the occurrence of clotting in deep veins; comparison to the time until clotting occurs in the heart cavities

Confirmation of the usefulness of the ultrasound-detected clotting in deep veins during resuscitation in assessing the severity of cardiac arrest and the prognosis of resuscitation, which is the aim of the project, will have an impact on international guidelines for determining the prognosis and potential futility of resuscitation.

DETAILED DESCRIPTION:
Introduction:

More than one million sudden cardiac arrests requiring cardiopulmonary resuscitation (CPR) occur each year in the United States and Europe. A point-of-care test to assess prognosis during resuscitation is a desirable clinical tool. Post-mortem intravascular clotting is considered an early sign of death. The detection of signs of clotting (spontaneous echo contrast or thrombus) in the cardiac cavities in an ultrasound examination during resuscitation may be an indicator of the severity of cardiac arrest and a marker of futile resuscitation. Performing transthoracic echocardiography during resuscitation is only possible during short breaks to assess the heart rhythm and pulse. Research shows that the use of transthoracic examination might cause additional interruptions in chest compressions. The use of a transesophageal examination, which can be performed during compressions, is only possible in specialized centers.

An examination that allows for the detection of intravascular clotting and at the same time does not require interruption of chest compressions is ultrasound assessment of deep veins. There is no data in the literature on the time that must pass from cardiac arrest to the occurrence of intravascular clotting, the frequency of clotting in deep veins during resuscitation and its importance for the resuscitation outcome.

Confirmation of the usefulness of the ultrasound-detected clotting in deep veins during resuscitation in assessing the severity of cardiac arrest and the prognosis of resuscitation, which is the aim of the project, will have an impact on international guidelines for determining the prognosis and potential futility of resuscitation.

Objectives of the study:

1. ultrasound assessment of the incidence of clotting in deep veins in patients after cardiac arrest during resuscitation and after the declaration of death; comparison to the incidence of clotting in the heart cavities
2. comparison of resuscitation results in patients with and without clotting detected in deep veins during resuscitation
3. determining the time from cardiac arrest to the occurrence of clotting in deep veins; comparison to the time until clotting occurs in the heart cavities

Methodology:

The study is planned to be prospective and double-blind. The study concerns emergency department patients after cardiac arrest who will undergo ultrasound examination during resuscitation and after declaration of death in the event of unsuccessful resuscitation. The first phase of the study will involve obtaining ultrasound images by clinicians not directly involved in patient care and resuscitation. Treating clinicians will be blinded to sonographic results except those concerning the cause of cardiac arrest. The images will then be externally evaluated for the presence of clotting by 2-3 assessors. These ultrasound assessors will be blinded to clinical outcomes of resuscitation and the timing of ultrasound examinations. The results of ultrasound examinations will be compared with data from the course and result of resuscitation. The time it takes for clotting to occur in the deep veins and heart cavities after cardiac arrest will also be determined.

The project concerns patients who suffered cardiac arrest and underwent cardiopulmonary resuscitation in the emergency department. The planned research group is 40 patients.

Timing of the ultrasound assessment Assessment of clotting in the deep veins and cardiac cavities during resuscitation will be performed once in every subsequent ten minutes of resuscitation (first examination: 1-10 minute of CPR; second examination: 11-20 minute of CPR, etc.). Bilateral ultrasound assessment of the common femoral veins and internal jugular veins will be performed during chest compressions, and transthoracic ultrasound assessment of the heart during breaks between chest compressions.

Assessment of clotting in the deep veins and heart cavities will be performed in three consecutive ten-minute periods after declaration of death (first examination: 1-10 minute; second examination: 11-20 minute; third examination 21-30 minute). The assessment will consist of bilateral ultrasound examination of the common femoral veins, internal jugular veins and transthoracic examination of the heart.

Study definitions Clotting will be considered present if the ultrasound image shows spontaneous echo contrast or thrombus.

Ultrasound protocols Ultrasound images will be obtained by the experts in point-of-care ultrasound who will not be directly involved in patient care and resuscitation. Each expert will be trained in the required examination protocol, including the time, type and quality of ultrasound examinations to be performed. Treating clinicians will be blinded to sonographic results to eliminate the risk of confounding from self-fulfilling prophecy. However, they will be informed of ultarsound findings that could influence clinical treatment such as mechanical ventricular activity and evidences of pulseless electrical activity reversible causes (pericardial effusion, right ventricular dilation, deep venous thrombosis in common femoral veins).

Ultrasonography imaging protocols followed during cardiac arrest and after declaration of death to assess clotting in the common femoral veins will rely on bilateral B-mode inspection for clotting and the compression ultrasound technique of the common femoral vein from the inguinal ligament until it becomes the femoral vein. Veins will be evaluated both in the transverse and longitudinal plane.

The protocols to assess clotting in the internal jugular veins will rely on bilateral B-mode inspection for clotting and the compression ultrasound technique of the internal jugular vein at three levels: (1) proximal portion of the jugular vein and the subclavian/innominate vein, (2) level of thyroid gland, (3) level of carotid bifurcation. Veins will be evaluated both in the transverse and longitudinal plane.

Echocardiography imaging protocols followed during cardiac arrest and after declaration of death will rely on three equivalent transthoracic B-mode views: (1) subcostal long-axis; (2) parasternal long-axis, (3) parasternal short-axis, and at minimum, (4) apical 4-chamber to assess all chambers for clotting.

The linear type of transducer will be used for the inspection of veins and the phased array type of transducer will be used for echocardiography.

Image adjudication All study images will be reviewed by at least 2 of 3 experts in point-of-care ultrasound to calculate inter-rater reliability for thrombus and spontaneous echo contrast identification. If there will be disagreement between diagnoses, a third reviewer would make the tiebreaker decision. These ultrasound assessors will be blinded to clinical outcomes of resuscitation and the timing of ultrasound examinations during the quality assurance oversight process.

Resuscitation data collection Other relevant resuscitation data concerning patient, pre-event data, cardiac arrest process and outcomes will be collected using the Utstein resuscitation registry template.

Potential Outcomes:

Confirmation of the usefulness of the ultrasound-detected clotting in deep veins during resuscitation in assessing the severity of cardiac arrest and the prognosis of resuscitation will have an impact on international guidelines for determining the prognosis and potential futility of resuscitation. Given the global number of cardiac arrests and resuscitations, shortening resuscitation efforts in selected cases will mean enormous savings in manpower and resources.

Confirmation of the effectiveness of the use of ultrasound in the assessment of early post-mortem changes in the vascular system may influence the development of forensic medicine through wider use of ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* patients who experience cardiac arrest in the emergency department, regardless of the mechanism and cause
* patients who were declared dead after resuscitation after cardiac arrest that occurred in the emergency department

Exclusion Criteria:

* age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who experience cardiac arrest in the emergency department, regardless of the mechanism and cause. Patients who were declared dead after resuscitation after cardiac arrest that occurred in the emergency department
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Intravascular clotting during CPR | One year (preliminary data will be presented after 6 months.
  The percentage of patients with intravascular clotting observed during cardioplumonary resuscitation.
Intravascular clotting after termination of CPR | One year (preliminary data will be presented after 6 months.
  The percentage of patients with intravascular clotting observed after termination of CPR
Time from cardiac arrest to first clot during CPR | One year (preliminary data will be presented after 6 months.
  Time from cardiac arrest to the first intravascular clot fromation during CPR
Time from cardiac arrest to first clot after termination of CPR. | One year (preliminary data will be presented after 6 months.
  Time from cardiac arrest to the first intravascular clot fromation after termination of CPR.

CONTACTS AND LOCATIONS:
Overall Officials: Robert K Szymczak, Asst. Prof., Principal Investigator — Medical University of Gdansk, Department of Emergency Medicine
Locations (1):
- University Clinical Centre - Clinical Emergency Department, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reynolds JC, Issa MS, C Nicholson T, Drennan IR, Berg KM, O'Neil BJ, Welsford M; Advanced Life Support Task Force of the International Liaison Committee on Resuscitation. Prognostication with point-of-care echocardiography during cardiac arrest: A systematic review. Resuscitation. 2020 Jul;152:56-68. doi: 10.1016/j.resuscitation.2020.05.004. Epub 2020 May 11. PMID 32437781
- [Background] Jackowski C, Thali M, Aghayev E, Yen K, Sonnenschein M, Zwygart K, Dirnhofer R, Vock P. Postmortem imaging of blood and its characteristics using MSCT and MRI. Int J Legal Med. 2006 Jul;120(4):233-40. doi: 10.1007/s00414-005-0023-4. Epub 2005 Nov 19. PMID 16328426
- [Background] Lau V, Blaszak M, Lam J, German M, Myslik F. Point-of-Care Resuscitative Echocardiography Diagnosis of Intracardiac Thrombus during cardiac arrest (PREDICT Study): A retrospective, observational cohort study. Resusc Plus. 2022 Mar 11;10:100218. doi: 10.1016/j.resplu.2022.100218. eCollection 2022 Jun. PMID 35299826
- [Background] Clattenburg EJ, Wroe P, Brown S, Gardner K, Losonczy L, Singh A, Nagdev A. Point-of-care ultrasound use in patients with cardiac arrest is associated prolonged cardiopulmonary resuscitation pauses: A prospective cohort study. Resuscitation. 2018 Jan;122:65-68. doi: 10.1016/j.resuscitation.2017.11.056. Epub 2017 Nov 23. PMID 29175356
- [Background] Scerrati A, Menegatti E, Zamboni M, Malagoni AM, Tessari M, Galeotti R, Zamboni P. Internal Jugular Vein Thrombosis: Etiology, Symptomatology, Diagnosis and Current Treatment. Diagnostics (Basel). 2021 Feb 23;11(2):378. doi: 10.3390/diagnostics11020378. PMID 33672254
- [Background] Nolan JP, Berg RA, Andersen LW, Bhanji F, Chan PS, Donnino MW, Lim SH, Ma MH, Nadkarni VM, Starks MA, Perkins GD, Morley PT, Soar J; Utstein Collaborators. Cardiac Arrest and Cardiopulmonary Resuscitation Outcome Reports: Update of the Utstein Resuscitation Registry Template for In-Hospital Cardiac Arrest: A Consensus Report From a Task Force of the International Liaison Committee on Resuscitation (American Heart Association, European Resuscitation Council, Australian and New Zealand Council on Resuscitation, Heart and Stroke Foundation of Canada, InterAmerican Heart Foundation, Resuscitation Council of Southern Africa, Resuscitation Council of Asia). Resuscitation. 2019 Nov;144:166-177. doi: 10.1016/j.resuscitation.2019.08.021. Epub 2019 Sep 16. PMID 31536777